CLINICAL TRIAL: NCT00557375
Title: Treatment Satisfaction Survey for Brain Tumor Patients and Their Caregivers
Brief Title: Brain Tumor Treatment Satisfaction Survey
Status: Completed | Type: Observational
Sponsor: Methodist Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: MHIRB 2007-036
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Brain Tumors
Keywords: Brain Tumors; Survey
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Brain tumor patients
- 2: Caregivers of brain tumor patients

SUMMARY:
Patients with recent diagnosis and treatment of a brain tumor will complete a short questionnaire concerning the patient's quality of life and emotional state since receiving treatment. Caregivers will complete a one-page questionnaire concerning the patient's quality of life and emotional state since receiving treatment.

DETAILED DESCRIPTION:
Patients with a recent diagnosis and treatment of a brain tumor (primary or metastatic; N=105, 61% female, 39% male) were identified in the clinics of Semmes-Murphey Neurologic and Spine Institute or the Methodist University Hospital in Memphis, TN. Caregivers were recruited from among relatives and friends who provide the most day-to-day care to the patient. All participants were between 3 months and 1 year from their most recent brain tumor treatment. Participants were given a simple, 5-point based survey to asses treatment-specific satisfaction, patient education, posttreatment quality of life, and pre- and post-treatment emotional impact. Therapeutic modalities surveyed include: surgery, external beam radiotherapy, whole-brain radiotherapy, stereotactic radiosurgery, and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are between 3 months and one year out from treatment for their brain tumor
* Karnofsky Performance Status (KPS) >= 60
* Age 18 years or over, any gender, any race
* "patient caregivers will be individuals who provide the most day-to-day care for their respective brain tumor patients

Exclusion Criteria:

* No exclusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Brain tumor patients and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2009-03-01 (Actual); Study Completion 2009-03-01 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction and emotional impact of treatments in patients who have undergone therapy(s)for brain tumors. | (greater than or equal to 3 months) from first treatment for brain tumor

SECONDARY OUTCOMES:
Observational data about the treatment course and emotional well-being of the brain tumor patient as provided by the caregiver. | (Greater than or equal to 3 months) from first treatment for brain tumor

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Sorenson, MD, Principal Investigator — Methodist Healthcare
Locations (1):
- Methodist University Hospital, Memphis, Tennessee, United States